CLINICAL TRIAL: NCT00202449
Title: A Placebo-Controlled Trial of Prazosin vs. Paroxetine in Combat Stress-Related PTSD Nightmares and Sleep Disturbance
Brief Title: Prazosin vs Paroxetine in Combat Stress-Related Post-Traumatic Stress Disorder (PTSD) Nightmares & Sleep Disturbance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Raskind 0046; DoD #PR054292 (Other Grant/Funding Number: Department of Defense); UW HS #04-1469-V 02 (Other: University of Washington)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Stress Disorders, Post-Traumatic; Sleep Disorders
Keywords: Prazosin; Paroxetine; Stress Disorders, Post-Traumatic; Sleep Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders | interventions — Prazosin; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Prazosin
  Interventions: Drug: prazosin
- 2 (Active Comparator): Paroxetine
  Interventions: Drug: paroxetine
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: prazosin — taken by mouth, twice daily, titrated up to efficacy or a maximum of 5 mg at 10a and 25 mg at bedtime for duration of study
  Other Names: Minipress
  Arms: 1
Drug: paroxetine — 20 mg taken at 10a for duration of the study
  Other Names: Paxil, Paxil CR
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The purposes of this study are:

* to evaluate the efficacy and tolerability of the drug prazosin compared to placebo for combat stress-related nightmares, sleep disturbance and overall function in recently combat-exposed returnees from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF).
* to evaluate the effects of the selective serotonin reuptake inhibitor (SSRI) paroxetine on behavioral symptoms and overall function in this population.

DETAILED DESCRIPTION:
Trauma-related nightmares and sleep disruption that follow combat exposure are distressing and frequently treatment resistant symptoms that impair quality of life and overall function. These symptoms closely resemble core nighttime symptoms of posttraumatic stress disorder (PTSD), and are increasingly recognized in returnees from Operation Iraqi Freedom (OIF) and Operation Enduring Freedom (OEF). Prazosin, a generically available brain active alpha-1 adrenergic receptor antagonist, markedly reduced or eliminated combat trauma-related nightmares and sleep disruption in 23 of 25 combat-exposed returnees from OIF at Madigan Army Medical Center (MAMC). The use of prazosin in OIF returnees was based on clinical efficacy of prazosin for trauma-related nightmares, sleep disturbance, and overall function in Vietnam combat veterans with chronic PTSD. The only drugs FDA approved for PTSD are the selective serotonin reuptake inhibitors (SSRIs) sertraline and paroxetine. However, SSRI effectiveness in combat trauma PTSD, especially for nighttime symptoms, remains questionable.

This is a placebo-controlled clinical trial of prazosin vs. the SSRI paroxetine for combat trauma-related nightmares, sleep disturbance, and overall posttraumatic stress disorder (PTSD) clinical severity in OIF/OEF returnees. Both neurobiologic considerations and our preliminary clinical treatment data provide support for the proposed trial. Preclinical and clinical studies suggest a role for increased central nervous system (CNS) adrenergic outflow and/or responsiveness in PTSD pathophysiology. Possible mechanisms include alpha-1 adrenergic receptor-mediated effects on sleep physiology, corticotropin releasing hormone secretion, and disruption of cognitive processing.

Here we propose a double-blind, placebo-controlled parallel group 12 week clinical trial of prazosin vs. paroxetine to test the following hypotheses:

Hypothesis 1. Prazosin will be more effective than paroxetine or placebo for reducing frequency and intensity of combat trauma-related nightmares (as measured by the "distressing dreams" item of the Clinician Administered PTSD Scale [CAPS]).

Hypothesis 2. Prazosin will be more effective than paroxetine or placebo for improving sleep quality (as measured by the Pittsburgh Sleep Quality Index [PSQI]).

Hypothesis 3. Prazosin will be more effective than paroxetine or placebo for improving overall clinical status (as measured by the Clinical Global Impression of Change [CGIC]).

Hypothesis 4. Prazosin will be better tolerated than paroxetine as measured by days retained in the study and frequency of adverse events.

Primary outcome measures will assess trauma-related nightmares, sleep disturbance and change in global clinical status: these will include the CAPS [59] Recurrent Distressing Dreams item, the PSQI (60) and the CGIC (58) score. Secondary outcome measures will include total CAPS score, the CAPS subscale scores (Reexperiencing/ Intrusions, Avoidance/Numbing, and Hyperarousal), the Nightmare Frequency Questionnaire (NFQ), Insomnia Severity Index, and measures of depressive signs and symptoms, quality of life, and number of study days completed.

ELIGIBILITY:
Inclusion Criteria:

* Hazardous duty in Iraq or Afghanistan with the US Armed Forces during Operations Iraqi Freedom and Operation Enduring Freedom
* Exposure to at least a moderate level of combat (>5 on Revised Combat Exposure Scale)
* Good general medical health
* Stable dose of non-excluded medications for at least 4 weeks prior to randomization
* >5 on CAPS recurrent distressing dreams item
* >5 on CAPS difficulty falling or staying asleep item

Exclusion Criteria:

* Acute or significant chronic medical illness, preexisting hypotension or orthostatic hypotension, pancreatitis, gout, Ménière's disease, benign positional vertigo, narcolepsy, or any other unstable medical condition.
* Women of childbearing potential with either positive pregnancy test or refusal to use effective birth control method will be excluded.
* Lifetime schizophrenia, schizoaffective disorder, bipolar disorder, psychotic disorder or any Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) cognitive disorder, current delirium, substance dependence disorder within 3 months of the study, severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others.
* Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist or paroxetine or any other SSRI, no concurrent use of another alpha-1 antagonist agent, no concurrent use of an antidepressant (other than trazodone prescribed for sleep).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray Raskind, MD, Principal Investigator — Director, Mental Health Services and Director, Mental Illness Research, Education, and Clinical Center VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Madigan Army Medical Center, Fort Lewis, Washington

REFERENCES:
- [Background] Raskind MA, Peskind ER, Kanter ED, Petrie EC, Radant A, Thompson CE, Dobie DJ, Hoff D, Rein RJ, Straits-Troster K, Thomas RG, McFall MM. Reduction of nightmares and other PTSD symptoms in combat veterans by prazosin: a placebo-controlled study. Am J Psychiatry. 2003 Feb;160(2):371-3. doi: 10.1176/appi.ajp.160.2.371. PMID 12562588
- [Background] Raskind MA, Thompson C, Petrie EC, Dobie DJ, Rein RJ, Hoff DJ, McFall ME, Peskind ER. Prazosin reduces nightmares in combat veterans with posttraumatic stress disorder. J Clin Psychiatry. 2002 Jul;63(7):565-8. doi: 10.4088/jcp.v63n0705. PMID 12143911
- [Background] Raskind MA, Dobie DJ, Kanter ED, Petrie EC, Thompson CE, Peskind ER. The alpha1-adrenergic antagonist prazosin ameliorates combat trauma nightmares in veterans with posttraumatic stress disorder: a report of 4 cases. J Clin Psychiatry. 2000 Feb;61(2):129-33. doi: 10.4088/jcp.v61n0208. PMID 10732660
- [Background] Peskind ER, Bonner LT, Hoff DJ, Raskind MA. Prazosin reduces trauma-related nightmares in older men with chronic posttraumatic stress disorder. J Geriatr Psychiatry Neurol. 2003 Sep;16(3):165-71. doi: 10.1177/0891988703256050. PMID 12967060

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin: Prazosin is a brain active alpha-1 adrenal receptor antagonist. Dose initiated at an initial dose of 1 mg qhs and titrated up to a maximum dose of 30 mg/day according to weight, age and presence or absence of daytime symptoms.
- Paroxetine: Paroxetine is a Selective Serotonin Reuptake Inhibitor. Dose started and maintained at 20 mg q10A.
- Placebo: Placebo is an inert substance used as a standard comparator in clinical pharmacologic trials.
Period: Overall Study
Arm/Group | Prazosin | Paroxetine | Placebo
Started | 18 | 20 | 21
Completed | 7 | 9 | 9
Not Completed | 11 | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Paroxetine | Placebo | Total
Number analyzed (Participants) | 18 | 20 | 21 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 21 | 59
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (7) | 28 (5) | 32 (9) | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 17 | 19 | 20 | 56
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 21 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Combat Trauma-related Nightmares From the Clinician Administered PTSD Scale (CAPS) Recurrent Distressing Dreams Item at Week 12
Description: Item B-2 "recurrent distressing dreams of the event" is a single item from the Clinician Administered PTSD Scale. The rating consists of two parts: Frequency and Intensity. Symptom frequency rated 0 to 4. Symptom intensity rated 0 to 4. Frequency plus Intensity ratings equal the total score. A higher score is worse; a lower score is better. This outcome measure evaluates the change in score from Baseline to Week 12. Minimum = 0 Maximum = 8
Time Frame: Baseline and Week 12
Population: Number of subjects analyzed equals the number of subjects who were able to complete this assessment at week 12 (e.g., completed the study).
Measure: Mean (Standard Deviation); unit: scale points
Arm/Group | Prazosin | Paroxetine | Placebo
Number analyzed (Participants) | 9 | 7 | 9
scale points | -1.29 (1.11) | -3.11 (2.52) | -2.67 (3.0)

2. Primary Outcome: Change in Sleep From the Pittsburgh Sleep Quality Index From Baseline to Week 12
Description: Pittsburgh Sleep Quality Index is a self-report questionnaire assessing sleep quality and disturbances over a 1-month time interval. A global score is obtained by summing the seven component subscales (total score range: 0-21). A score of 5 or less indicates good sleep quality. A score of more than 5 indicates poor sleep quality. Change is measured from Baseline to Week 12.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scale points
Arm/Group | Prazosin | Paroxetine | Placebo
Number analyzed (Participants) | 6 | 9 | 9
scale points | -2.33 (2.94) | -6.44 (3.91) | -3.33 (5.45)

3. Primary Outcome: Change in Global Trauma-related Symptom Severity and Functioning From the Clinical Global Impression of Change From Baseline to Week 12
Description: The Clinical Global Impression of Change is a 7-point scale that rates global change compared to baseline (1=markedly improved, 2=moderately improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=moderately worse, 7=markedly worse). The CGIC is used to determine the impact of treatment effects on meaningful and distinct change in overall sense of well-being and functioning. This outcome measure evaluates change from baseline to Week 12.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scale points
Arm/Group | Prazosin | Paroxetine | Placebo
Number analyzed (Participants) | 7 | 9 | 9
scale points | 3.14 (1.86) | 2.11 (1.05) | 2.33 (1.22)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events were collected over the course of 12 weeks.
Arm/Group | Prazosin | Paroxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 3/18 | 3/20 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=18) | Paroxetine (N=20) | Placebo (N=21)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
dry mouth (General disorders) | 0 (0) | 0 (0) | 1 (1)
dizziness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
numbness in face and hands (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
heart palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
anxiety with palpitations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
allertic reaction to tramadol - hives/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAK bilateral eye surgery (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
nocturnal urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
panic attack (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
change in vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
central chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
reaction to study drug (paroxetine) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
abnormal ejaculation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
difficulty concentrating (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
surgery for dyskinesia of esophagus and diverticulum of esophagus, acquired. (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
High rate of early termination leading to small number of patients analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No